CLINICAL TRIAL: NCT03227588
Title: Evaluation of the Opsens Fractional Flow Reserve (FFR) Wire as a "Work Horse" Wire
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Uretsky, Director of Interventional Cardiology and Cath Lab, Central Arkansas Veterans Healthcare System
Other Study IDs: 966635
Record Dates: First submitted 2017-06-27; First posted 2017-07-24 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fractional Flow Reserve — This is a prospective data collection study for patients that have undergone FFR.

SUMMARY:
The use of fractional flow reserve (FFR) has improved outcomes in percutaneous coronary interventions (PCI) in patients with symptomatic stable coronary artery disease (CAD) with intermediate angiographic stenoses. It is a clinical tool used routinely in cardiac catheterization laboratories throughout the world including the Little Rock VA Hospital. The technique utilizes a pressure transducer constructed as part of an 0.014" guidewire. An FFR of >0.80 has been linked with myocardial ischemia found with nuclear stress and dobutamine echo stress testing. The FAME trial clearly demonstrated its value in improving long-term outcomes as compared to use of angiography alone. As such, the use of FFR is incorporated into both AHA ACC and European PCI guideline recommendations as part of routine care for intermediate lesions. A "work horse" guide wire is so defined because it can be used in most PCI cases. It combines a low tip load (to avoid intimal dissection, with excellent (ideally, one to one) torque transmission and trackability through tortuous lesions. Recently the FDA has approved an FFR guide wire, OptoWire, (Opsens, Quebec City, Quebec, CAN) which uses light transmission to measure pressure rather than electrical transduction wires. The primary purpose of the present study is to determine how effective this wire is as a work horse wire in patients in whom FFR is required. The OptoWire may also have the advantage of less "drift" occurring during the procedure. Drift refers to the change in pressure due to issues related to the wire and measuring system, rather than a true change in pressure. All current FFR wire systems demonstrate some degree of drift requiring measuring pressure of the wire in the aorta after the procedure is completed to determine if, and to what extent, drift has occurred. Thus, a secondary aim of this study will determine the degree of drift.

DETAILED DESCRIPTION:
EVALUATION OF THE OPSENS FRACTIONAL FLOW RESERVE (FFR) WIRE AS A "WORK HORSE" WIRE

INVESTIGATORS:

PRINCIPAL INVESTIGATOR: BARRY F URETSKY, MD CO-INVESTIGATOR: ABDUL HAKEEM, MD CO-INVESTIGATOR: MALEK AL-HAWWAS, MD

Introduction The use of fractional flow reserve (FFR) has improved outcomes in percutaneous coronary interventions (PCI) in patients with symptomatic stable coronary artery disease (CAD) with intermediate angiographic stenoses. It is a clinical tool used routinely in cardiac catheterization laboratories throughout the world including the Little Rock VA hospital. The technique utilizes a pressure transducer constructed as part of an 0.014" guidewire. The wire is passed distal to the stenosis. Under the condition of maximal hyperemia induced by a drug, typically adenosine, the pressure proximal to the stenosis, i.e. aortic pressure or Pa and the pressure distal to the stenosis, Pd, are measured. The ratio, Pd/Pa, under maximal flow or hyperemia is known as the fractional flow reserve (FFR). An FFR of <0.80 has been correlated with observed myocardial ischemia using other diagnostic methods, particularly nuclear stress and dobutamine echo stress testing. The FAME trial clearly demonstrated its value in improving long-term outcomes as compared to use of angiography alone (1). As such, the use of FFR is incorporated into both AHA ACC and European PCI guideline recommendations as part of routine care for intermediate lesions (2,3).

One of the limitations of the use of the FFR pressure wire itself is that its handling characteristics are somewhat inferior to a standard "work horse" guide wire used for PCI. A "work horse" guide wire is so defined because it can be used in most PCI cases. It combines a low tip load (to avoid intimal dissection) with excellent (ideally, one-to-one) torque transmission and trackability through tortuous lesions. There are several different work horse wires available. Although the wires may be different for different Cath Labs and operators, the wires are universally used to maximize safety, efficacy, and efficiency of PCI.

In patients specifically requiring FFR to determine the value of PCI, it would be ideal if an FFR wire was as effective as a work horse wire so it could be used in difficult-to-traverse lesions. However, due to the complex electronics within current FFR wires, handling characteristics of previously used wires are inferior to current work horse wires. Recently the FDA has approved an FFR guide wire, OptoWire, (Opsens, Quebec City, Quebec, CAN) using light transmission to measure pressure rather than electrical transduction (4). It is commercially available in the United States. Its handling characteristics appear to approach that of a work horse guide wire and may represent an improvement over electrical transduction wires. The primary purpose of the present study is to determine how effective this wire is as a work horse wire in patients in whom FFR is required.

The OptoWire may also have the advantage of less "drift" occuring during the procedure. Drift refers to the change in pressure due to issues related to the wire and measuring system, rather than a true change in pressure. All current FFR wire systems demonstrate some degree of drift requiring measuring pressure of the wire in the aorta after the procedure is completed to determine if, and to what extent, drift has occurred. Thus, a secondary aim of this study will determine the degree of drift.

In clinical practice, FFR is performed before, and often after, PCI. In a study of 574 patients treated at the Little Rock VA (IRB Study, #779601), teh investigators found that approximately 20% of angiographically optimized PCI still had an ischemic FFR. The investigators further found that this ischemic value could be improved by further treatments including balloon angioplasty and stenting. Thus, the secondary purpose is to measure FFR after successful PCI to ascertain the incidence of persistently ischemic FFR after optimized angiographic stenting to confirm the result from out previous study.

Statistical analysis

This study is descriptive. It will use means and standard deviation for continuous variables and prevalence or incidence in percentages as appropriate to show results. As there is no comparator group, comparative statistics will not be employed.

Research aspect of study

The research aspect of the study is limited to the systematic collection and analysis of data using the Opsens FFR wire with plan for publication. The other aspects of the study are considered part of routine clinical care. They include passage of FFR wire, measurement of FFR pre- and post-PCI, and performance of PCI itself.

Significance of study

A wire that can be used as a workhorse as well as be able to measure FFR would be of great value. The more effective and efficient is the FFR wire in not only measuring pre-PCI FFR but being able to be used for PCI and be stable and durable enough to be used for post-PCI optimization, the greater is the probability that this approach will be more generally adopted into clinical practice. Demonstration that the Opsens FFR wire is effective in this regard should further this goal.

The investigators previously demonstrated that 21% or about 1 in 5 patients had an ischemic FFR after satisfactory angiographic result. This study will confirm previous results or suggest either an over- or under-estimation of that incidence.

ELIGIBILITY:
Inclusion Criteria:

Patients (age 18-89 years old) eligible and in whom the operator has performed FFR will be included to systematically evaluate the performance of the OptoWire FFR wire. A total of 1000 consecutive patients deemed to require FFR as part of clinical care will be included. It is felt that 1000 patients represent a reasonable sample size to study the OptoWire FFR wire handling characteristics, the primary endpoint of the study

Exclusion Criteria:

1. Not a candidate for FFR
2. Chronic total occlusion lesion
3. Hemodynamically unstable
4. Saphenous vein graft lesions -

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (age 18-89 years old) eligible and in whom the operator has performed FFR will be included to systematically evaluate the performance of the OptoWire FFR wire. A total of 1000 consecutive patients deemed to require FFR as part of clinical care will be included. It is felt that 1000 patients represent a reasonable sample size to study the OptoWire FFR wire handling characteristics, the primary endpoint of the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-12-10 (Estimated); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
Opsens FFR Wire Performance | Acute result at end of procedure
  Satisfactory performance is defined as the ability to perform the entire PCI plus measure FFR pre and post PCI with drift <0.05.

SECONDARY OUTCOMES:
Incidence of Ischemic or Low Non-ischemic FFR post PCI requiring further intervention | Acute result at end of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Barry F. Uretsky, MD, Principal Investigator — CAVHS
Locations (1):
- John L. McClellan Memorial Veterans Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Costa F, Ariotti S, Valgimigli M, Kolh P, Windecker S; Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Perspectives on the 2014 ESC/EACTS Guidelines on Myocardial Revascularization : Fifty Years of Revascularization: Where Are We and Where Are We Heading? J Cardiovasc Transl Res. 2015 Jun;8(4):211-20. doi: 10.1007/s12265-015-9632-6. Epub 2015 May 19. PMID 25986910
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Society for Cardiovascular Angiography and Interventions. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. J Am Coll Cardiol. 2011 Dec 6;58(24):e44-122. doi: 10.1016/j.jacc.2011.08.007. Epub 2011 Nov 7. No abstract available. PMID 22070834
- [Background] Agarwal SK, Kasula S, Hacioglu Y, Ahmed Z, Uretsky BF, Hakeem A. Utilizing Post-Intervention Fractional Flow Reserve to Optimize Acute Results and the Relationship to Long-Term Outcomes. JACC Cardiovasc Interv. 2016 May 23;9(10):1022-31. doi: 10.1016/j.jcin.2016.01.046. PMID 27198682
- [Derived] Uretsky BF, Agarwal SK, Vallurupalli S, Al-Hawwas M, Hasan R, Miller K, Hakeem A. Prospective Evaluation of the Strategy of Functionally Optimized Coronary Intervention. J Am Heart Assoc. 2020 Feb 4;9(3):e015073. doi: 10.1161/JAHA.119.015073. Epub 2020 Jan 30. PMID 32013707
- See also: Optowire product information — http://opsensmedical.com/products/optowire/